CLINICAL TRIAL: NCT03460106
Title: The Development of a Screening Assay by LC-MS/MS to Monitor Adherence to Asthma Treatment
Acronym: SALMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart of England NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2017097RM
Record Dates: First submitted 2018-02-23; First posted 2018-03-09 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: Asthma Medical Adherence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Phase I: To develop and validate laboratory urine and blood test for the detection of medications commonly used in the treatment of asthma Phase II: to test the developed assay in the clinic, to determine its practicality to conduct, and its clinical utility in adherence assessment.

DETAILED DESCRIPTION:
Phase I: laboratory based study to develop LC-MS/MS assay of urine / blood to detect presence or lack asthma medication in 50 volunteers with asthma. Phase II: once the test is validated it will be tested in a 100 patients attending the asthma clinics to test its clinical utility. Urine and blood samples will be collected from patients at time of clinic attendance to test for asthma medication panel and outcome will determine adherence or non-adherence. Clinical outcomes of adherent versus non adherent groups will be compared in terms of asthma control, lung function, biomarkers FeNO and blood eosinophils, exacerbation frequency and hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80
2. Able to give valid informed consent
3. Prescribed one or more of the medications to be tested
4. Able to provide a blood and urine sample
5. Able to complete questionnaires in English

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Patients known to have any blood borne virus that would render the sample hazardous. This includes Hepatitis B, Hepatitis C and HIV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified at the BRSAS, general asthma clinics and as inpatients admitted to wards at HEFT. The research team will approach patients in these settings.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
To develop and validate laboratory urine and blood test for the detection of medications commonly used in the treatment of asthma | 4 months
  5ml biochemistry SST and 2.5ml EDTA blood sample and urine 10ml sample will be collected simultaneously from the patient on the same day and transferred to biochemistry department at Heartlands hospital. These samples will be used to develop and validate the assays

SECONDARY OUTCOMES:
To test the developed assay in the clinic, to determine its practicality to conduct, and its clinical utility in adherence assessment. | 6 months
  Patients' assessment will be similar to that described in phase I, however in phase II the administration treatment will not be directly observed. Patients will be recruited from the clinic. Patients will be asked to identify the time they took their prescribed medication and asked to provide a 5ml biochemistry SST and 2.5ml EDTA blood sample and urine 10ml sample.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mr Williams, Principal Investigator — Heart of England NHS Foundation Trust; Alexander Lawson Dr Lawson, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Birmingham Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No